CLINICAL TRIAL: NCT00587457
Title: A Phase I, Multicenter, Dose-Escalation Study of CAT-8015 in Patients With Relapsed or Refactory Chronic Lymphocytic Leukemia (CLL) Prolymphocytic Leukemia (PLL), or Small Lymphocytic Leukemia (SLL)
Brief Title: A Phase I, Multicenter, Dose Escalation Study of CAT-8015 in Participants With Chronic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is terminated early due to unavailability of investigational product.
Sponsor: MedImmune LLC (Industry)
Collaborators: Cambridge Antibody Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-8015-1002
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Leukemia, Lymphoma, Chronic Lymphocytic; Leukemia, Prolymphocytic Leukemia, Small; Lymphocytic Lymphoma, Moxetumomab Pasudotox
Keywords: Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Small Lymphocytic Lymphoma; Moxetumomab pasudotox
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Prolymphocytic; Cerebral Palsy; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — immunotoxin HA22

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CAT-8015 5 microgram per kilogram (mcg/kg) (Experimental): Participants received a single intravenous infusion of 5 mcg/kg moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until progressive disease (PD) or until otherwise they become ineligible.
  Interventions: Drug: CAT-8015 5 mcg/kg
- CAT-8015 10 mcg/kg (Experimental): Participants received a single intravenous infusion of 10 mcg/kg moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until progressive disease (PD) or until otherwise they become ineligible.
  Interventions: Drug: CAT-8015 10 mcg/kg
- CAT-8015 20 mcg/kg (Experimental): Participants received a single intravenous infusion of 20 mcg/kg moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until progressive disease (PD) or until otherwise they become ineligible.
  Interventions: Drug: CAT-8015 20 mcg/kg

INTERVENTIONS:
Drug: CAT-8015 5 mcg/kg — Participants received a single intravenous infusion of 5 mcg/kg moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until progressive disease (PD) or until otherwise they become ineligible.
  Arms: CAT-8015 5 microgram per kilogram (mcg/kg)
Drug: CAT-8015 10 mcg/kg — Participants received a single intravenous infusion of 10 mcg/kg moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until progressive disease (PD) or until otherwise they become ineligible.
  Arms: CAT-8015 10 mcg/kg
Drug: CAT-8015 20 mcg/kg — Participants received a single intravenous infusion of 20 mcg/kg moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until progressive disease (PD) or until otherwise they become ineligible.
  Arms: CAT-8015 20 mcg/kg

SUMMARY:
This was a multicenter, Phase 1, standard 3+3 dose-escalation study to evaluate the safety and anti-neoplastic activity of moxetumomab pasudotox in relapsed or refractory participants with chronic lymphocytic leukemia (CLL), prolymphocytic leukemia (PLL) or Small Lymphocytic Lymphoma (SLL).

DETAILED DESCRIPTION:
This was a multicenter, Phase 1, standard 3+3 dose-escalation study to evaluate the safety and anti-neoplastic activity of CAT-8015 in relapsed or refractory participants with CLL, PLL, or SLL. Participants in the initial dose cohort were to receive CAT-8015 at a dose of 5 microgram per kilogram (mcg/kg) CAT-8015, increasing to 10 mcg/kg in the second dose cohort, and then increasing by 10 mcg/kg increments in subsequent cohorts (that is, to doses of 20, 30, 40, 50, 60 mcg/kg, etc) until a maximum tolerated dose (MTD) was identified. Following identification of the MTD, the MTD cohort was to be expanded to 16 participants.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of B-Cell Leukemia [(chronic lymphocytic leukemia (CLL), prolymphocytic leukemia (PLL), or Small lymphocytic leukemia (SLL)]
* Measurable Disease
* Disease characteristics: Participants with CLL or SLL are eligible if they have failed 2 or more prior courses of standard chemo and/or biologic therapy (example, Rituxan) and PLL will be eligible if they have failed at least one prior standard chemotherapeutic regimen. Medical indications for treatment include progressive disease-related symptoms, progressive cytopenias due to marrow involvement, progressive or painful splenomegaly or adenopathy, rapidly increasing lymphocytosis, autoimmune hemolytic anemia or thrombocytopenia and increased frequency of infections.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Participants with other cancers who meet eligibility criteria and have had less than 5 years of disease-free survival will be considered on a case-by-case basis
* Life expectancy of greater than 6 months, as assessed by the principal investigator
* Must be able to understand and sign the informed consent
* Must be at least 18 years old
* Female and Male participants agree to use an approved method of contraception during the study

Exclusion Criteria:

* History of allogeneic bone marrow transplant.
* Documented and ongoing central nervous system involvement with their malignant disease [history of central nervous system (CNS) involvement is not an exclusion criterion]
* Pregnant or breast-feeding females
* Participants who plasma contains either a significant level of antibody to CAT-8015 as measured by ELISA, or antibody that neutralizes the binding of CAT-8015 to CD22 as measured by a competition ELISA.
* HIV positive serology (due to increased risk of severe infection and unknown interaction of CAT-8015 with antiretroviral drugs)
* Hepatitis B surface antigen positive
* Uncontrolled, symptomatic, intercurrent illness including but not limited to: infections requiring systemic antibiotics, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements.
* Hepatic function: Serum transaminases [either alanine aminotransferase (ALT) or aspartate aminotransferase (AST)] or direct bilirubin greater than or equal to Grade 2, unless bilirubin is due to Gilbert's disease
* Renal function: Serum creatinine clearance is less than or equal to 60 millilitre per minute (mL/min) as estimated by Cockcroft-Gault formula

Hematologic function:

* The ANC less than 1000/cubic millimeter (cmm), or platelet count less than 50,000/cmm, if these cytopenias are not judged by the investigator to be due to underlying disease (that is, potentially reversible with anti-neoplastic therapy).
* A participant will not be excluded because of pancytopenia greater than or equal to Grade 3, or erythropoietin dependence, if it is due to disease, based on the results of bone marrow studies.
* Baseline coagulopathy greater than or equal to grade 3 unless due to anticoagulant therapy

Pulmonary function:

- Participants with less than 50 percent (%) of predicted forced expiratory volume (FEV-1) or less than 50% of predicted diffusing capacity for carbon monoxide (DLCO) corrected for hemoglobin concentration and alveolar volume. Note: Participants with no prior history of pulmonary illness are not required to have pulmonary function test (PFTs). FEV1 will be assessed after bronchodilator therapy.

Recent prior therapy:

* Cytotoxic chemotherapy, corticosteroids (except stable doses of prednisone), whole body electron beam radiation therapy, hormonal, biologic or other standard or any investigational therapy of the malignancy for 3 weeks prior to entry into the trial.
* Less than or equal to 1 month prior monoclonal antibody therapy (that is, rituximab)
* Participants who are receiving or have received radiation therapy less than 3 weeks prior to study entry will not be excluded providing the volume of the bone marrow treated is less than 10% and also the participant has measurable disease outside the radiation report.
* Any history of prior pseudomonas - exotoxin immunotoxin administrator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-03-07 (Actual); Primary Completion 2008-04-07 (Actual); Study Completion 2008-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Lanasa, M.D.,Ph.D, Study Director — MedImmune LLC
Locations (3):
- United States (2):
  - Research Site, Indianapolis, Indiana
  - Research Site, Bethesda, Maryland
- Research Site, Lodz, Poland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 11 participants were enrolled, of which all participants discontinued from the treatment.
Groups:
- CAT-8015 10 Microgram Per Kilogram (mcg/kg): Participants received a single intravenous infusion of 10 mcg/kg moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until progressive disease (PD) or until otherwise they become ineligible.
- CAT-8015 20 Microgram Per Kilogram (mcg/kg): Participants received a single intravenous infusion of 20 mcg/kg moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until progressive disease (PD) or until otherwise they become ineligible.
Period: Overall Study
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Started | 3 | 3 | 5
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 5
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Disease progression | 2 | 0 | 2
Not completed — Initiation of alternative therapy | 0 | 1 | 0
Not completed — Undefined | 0 | 0 | 1
Not completed — Development of neutralizing Abs | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg) | Total
Number analyzed (Participants) | 3 | 3 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (2.3) | 62.0 (4.4) | 61.6 (7.5) | 60.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 2 | 2 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) events present at baseline that worsened in intensity after administration of investigational product or events absent at baseline that emerged after administration of study drug, for the period extending to 30 days after the last dose of study drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening situation (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received moxetumomab pasudotox. Treatment-emergent were events between administration of investigational product and Day 28 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Number; unit: Participants
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
Participants
  TEAEs | 3 | 3 | 5
  TESAEs | 1 | 2 | 3

2. Primary Outcome: Number of Participants With Vital Signs Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: The vital sign abnormalities which require an action or intervention by the investigator, or a finding judged by the investigator were reported as an adverse event. TEAEs were events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug, for the period extending to 30 days after the last dose of study drug.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Number; unit: Participants
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
Participants
  Pyrexia | 1 (0.56) | 0 (0.70) | 1 (0.29)
  Sinus tachycardia | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Relevant Electrocardiogram (ECG) Abnormalities Recorded as Adverse Events (AEs)
Description: AEs observed in participants with clinically significant ECG abnormalities were assessed.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Number; unit: Participants
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Treatment-emergent were events between first dose of study drug and 30 days after the last dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with grade 3 or higher treatment-emergent adverse events for laboratory abnormalities were reported as clinically relevant laboratory changes.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Number; unit: Participants
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
Participants
  Hemoglobin decreased | 3 | 0 | 1
  Platelet count decreased | 2 | 1 | 1
  Neutrophil count decreased | 2 | 0 | 0
  Lymphocyte count decreased | 1 | 0 | 0
  White blood cell count decreased | 1 | 0 | 0
  Neutropenia | 1 | 0 | 0
  Febrile neutropenia | 0 | 1 | 0
  Blood albumin decreased | 1 | 1 | 2
  Blood magnesium decreased | 1 | 2 | 0
  Blood glucose increased | 2 | 0 | 0
  Blood magnesium increased | 1 | 1 | 0
  Blood phosphorus decreased | 1 | 1 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0
  Blood alkaline phosphatase increased | 0 | 1 | 0
  Blood calcium increased | 0 | 1 | 0
  Blood glucose decreased | 0 | 0 | 1
  Blood potassium decreased | 0 | 1 | 0
  Blood sodium decreased | 1 | 0 | 0
  Blood sodium increased | 0 | 1 | 0
  Blood triglycerides increased | 1 | 0 | 0

5. Primary Outcome: Number of Participants With Objective Response Rate (ORR): Complete Response (CR) or Partial Response (PR)
Description: Objective response rate defined as the proportion of participants with confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria.
Time Frame: Up to 2 years of post-treatment follow-up
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Number; unit: Participants
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
Participants | 0 | 0 | 0

6. Primary Outcome: Best Overall Objective Tumor Response
Description: Antitumor activity was assessed by best overall objective tumor response.
Time Frame: Up to 2 years of post-treatment follow-up
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Number; unit: Participants
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
Participants
  Complete response (CR) | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0
  Stable Disease (SD) | 2 | 3 | 2
  Progressive Disease (PD) | 1 | 0 | 3

7. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Moxetumomab Pasudotox
Description: The Tmax is the time to reach maximum observed plasma concentration of Moxetumomab Pasudotox.
Time Frame: Predose, 0.25 (During Infusion), 0.5 (End of Infusion), 1, 1.5, 2, 4, 8 and 12 hours postdose on Day 1 and 5; Predose and End of Infusion on Day 3
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox. Here 'n' signifies participants evaluable for specified categories, for each arm, respectively.
Measure: Median (Full Range); unit: hour
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
hour
  Cycle 1, Day 1 (n=3,3,5) | 0.500 [0.500 to 0.500] | 0.50 [0.500 to 0.500] | 0.500 [0.00 to 0.500]
  Cycle 1, Day 5 (n=3,3,5) | 0.500 [0.500 to 0.500] | 0.500 [0.300 to 0.500] | 0.500 [0.300 to 1.00]
  Cycle 2, Day 1 (n=2,2,2) | 4.25 [0.500 to 8.00] | 0.375 [0.250 to 0.500] | 0.500 [0.500 to 0.500]
  Cycle 2, Day 5 (n=2,2,2) | 0.500 [NA to NA] — Participant had no measurable Tmax concentration. | 0.800 [0.500 to 1.00] | 0.500 [0.500 to 0.500]
  Cycle 3, Day 1 (n=1,1,2) | 0.500 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | 0.500 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | 0.500 [0.500 to 0.500]
  Cycle 3, Day 5 (n=1,1,2) | 0.500 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | 2.00 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | 0.500 [0.500 to 0.500]
  Cycle 4, Day 1 (n=1,NA,NA) | 0.500 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 4, Day 5 (n=1,NA,NA) | 0.500 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 5, Day 1 (n=1,NA,NA) | 0.500 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 5, Day 5 (n=1,NA,NA) | 0.500 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 6, Day 1 (n=1,NA,NA) | 0.500 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 6, Day 5 (n=1,NA,NA) | 0.500 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.

8. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for Moxetumomab Pasudotox
Description: The Cmax is the maximum observed plasma concentration of Moxetumomab Pasudotox.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: nanogram per milliliter
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
nanogram per milliliter
  Cycle 1, Day 1 (n=3,3,5) | 97 [59.1 to 107] | 57.7 [46.5 to 145] | 180 [63.7 to 351]
  Cycle 1, Day 5 (n=3,3,5) | 80.9 [56.4 to 122] | 117 [44.7 to 166] | 206 [108 to 353]
  Cycle 2, Day 1 (n=2,2,2) | 94.0 [66.0 to 122] | 723 [146 to 1300] | 156 [134 to 178]
  Cycle 2, Day 5 (n=2,2,2) | 50.5 [0.00 to 101] | 80.8 [72.3 to 89.2] | 211 [171 to 250]
  Cycle 3, Day 1 (n=1,1,2) | 107 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | 154 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | 160 [63.9 to 257]
  Cycle 3, Day 5 (n=1,1,2) | 93.4 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | 200 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | 266 [156 to 376]
  Cycle 4, Day 1 (n=1,NA,NA) | 84.9 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 4, Day 5 (n=1,NA,NA) | 86.2 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 5, Day 1 (n=1,NA,NA) | 95.0 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 5, Day 5 (n=1,NA,NA) | 86.9 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 6, Day 1 (n=1,NA,NA) | 93.2 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.
  Cycle 6, Day 5 (n=1,NA,NA) | 67.0 [NA to NA] — Median range was not evaluable since only 1 participant was evaluated. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected. | NA [NA to NA] — Data was not evaluated due to the small size of the sample cohorts and limited quantifiable data collected.

9. Secondary Outcome: Number of Participants With Positive Neutralizing Antibodies
Description: Participants tested for immunogenicity to moxetumomab pasudotox prior to enrollment, before each cycle and at end of study. The neutralization assay measures the capacity of participant's plasma (antibodies) to inhibit the binding of moxetumomab pasudotox to its target, cluster of differentiation 22 (CD22), coated onto enzyme linked immunosorbent assay (ELISA) plates. It was used as a direct surrogate for biological activity based on the mechanism of action of this drug. Significant level of neutralizing antibody activity defined as the capacity of test plasma to inhibit greater than (>)50 percentage (%) of the binding of CAT-8015 to CD22 using an ELISA-based method.
Time Frame: Up to end of treatment (4-6 weeks after the last dose)
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Number; unit: Participants
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
Participants | 0 | 0 | 1

10. Secondary Outcome: Percentage Change From Baseline in Cluster of Differentiation 22 (CD22) Expression
Description: Participants demonstrated CD22 expression on malignant cells at Screening and CD22 is a regulatory molecule that prevents the over activation of the immune system and the development of autoimmune diseases.
Time Frame: End of treatment (4-6 weeks after the last dose)
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 3 | 3 | 5
Percentage
  CD22-PE [OF CD5+/CD19+] | -33.65 (27.79) | -10.25 (16.05) | -8.85 (16.19)
  (MESF CD22-PE [of CD5+/CD19+]) | 1139 (1514.6) | -3076 (5982.1) | -342.8 (1816.8)

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 30 days after the last dose of study drug
Arm/Group | CAT-8015 5 Microgram Per Kilogram (mcg/kg) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) | CAT-8015 20 Microgram Per Kilogram (mcg/kg)
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 3/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAT-8015 5 Microgram Per Kilogram (mcg/kg) (N=3) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) (N=3) | CAT-8015 20 Microgram Per Kilogram (mcg/kg) (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary histoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAT-8015 5 Microgram Per Kilogram (mcg/kg) (N=3) | CAT-8015 10 Microgram Per Kilogram (mcg/kg) (N=3) | CAT-8015 20 Microgram Per Kilogram (mcg/kg) (N=5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 1 (5) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (2) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Histoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 1 (2) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Blood magnesium increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 3 (6) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (3) | 1 (2) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (3) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to unavailability of investigational product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.